## Plantar Pressure Distribution in Relation to The Way of Carrying Backpack in Adolescentes

**⋄** NCT Number

NCT07161349

Date:

Sept-2023

## **Sample Consent Form**

| I am Freely and voluntarily consent to participate of |
|-------------------------------------------------------------------------|
| my child in this research study (PLANTAR PRESSURE DISTRIBUTION |
| IN RELATION TO THE WAY OF CARRYING BACKPACK IN |
| ADOLESCENTES) |
| Under the direction of researcher Amira Ibrahem Mohamed. |
| Description of the procedures has been explained to me and I understand |
| that I may withdraw my consent and discontinue participation in this |
| research at any time without prejudice to me. |
| Date: / / 20 |

Participant: .....